CLINICAL TRIAL: NCT00017043
Title: A Phase II Study of Epothilone Analog BMS-247550 in Patients With Metastatic Gastric Adenocarcinoma Previously Treated With a Taxane
Brief Title: BMS-247550 in Treating Patients With Metastatic Stomach Cancer Previously Treated With Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068644; BMS-MSKCC-01011; MSKCC-01011; NCI-G01-1949
Record Dates: First submitted 2001-06-06; First posted 2003-09-09 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: stage IV gastric cancer; recurrent gastric cancer; stage IV esophageal cancer; recurrent esophageal cancer; adenocarcinoma of the stomach; adenocarcinoma of the esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Adenocarcinoma Of Esophagus | interventions — ixabepilone

INTERVENTIONS:
Drug: ixabepilone

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of BMS-247550 in treating patients who have metastatic stomach cancer previously treated with chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the clinical activity of BMS-247550, in terms of response rate, in patients with previously treated metastatic gastric adenocarcinoma.
* Determine the safety of this drug in these patients.
* Assess the response duration, time to progression, and survival of patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive BMS-247550 IV over 1 hour on day 1. Treatment repeats every 21 days for 2-18 courses in the absence of disease progression or unacceptable toxicity. Patients with a complete response (CR) receive 4 additional courses after confirmation of CR.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 21-58 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma originating in the stomach or gastroesophageal junction

  * Failed prior taxane-based chemotherapy regimen* in the metastatic setting OR
  * Relapsed within 6 months of completing taxane-based chemotherapy* in the adjuvant setting
* Bidimensionally measurable metastatic disease

  * No prior radiotherapy to only measurable target lesion
* No squamous cell or sarcomatous disease
* No known brain metastases NOTE: *Regimen must have included a fluopyrimidine and/or a platinum drug

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Absolute neutrophil count at least 2,000/mm^3
* Platelet count greater than 125,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* ALT no greater than 2.5 times ULN (5 times ULN if liver metastases present)

Renal:

* Creatinine no greater than 2 times ULN

Cardiovascular:

* No unstable angina, myocardial infarction, or congestive heart failure within the past 6 months

Other:

* No other malignancy within the past 2 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No serious concurrent infection
* No nonmalignant uncontrolled medical illness that would preclude study
* No psychiatric disorder or other condition that would preclude study compliance
* No neuropathy (neuromotor or neurosensory) of grade 2 or greater
* No known severe hypersensitivity to agents containing Cremophor EL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 2 months after the study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent immunotherapy

Chemotherapy:

* See Disease Characteristics
* At least 3 weeks since prior chemotherapy for metastatic disease
* Prior neoadjuvant and adjuvant chemotherapy allowed
* No more than 1 prior chemotherapy regimen for metastatic disease
* No other concurrent chemotherapy

Endocrine therapy:

* No concurrent hormonal therapy except hormone replacement therapy

Radiotherapy:

* See Disease Characteristics
* At least 3 weeks since prior radiotherapy and recovered
* No prior radiotherapy to major bone marrow-containing areas (e.g., pelvis or lumbar spine)
* No concurrent therapeutic radiotherapy

Surgery:

* At least 1 week since prior minor surgery and recovered
* At least 3 weeks since prior major surgery and recovered

Other:

* No other concurrent experimental anticancer medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-02; Primary Completion 2003-01 (Actual); Study Completion 2003-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manish A. Shah, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States